CLINICAL TRIAL: NCT05627518
Title: A Randomized, Single Dose, Crossover Study in Healthy Volunteers to Investigate the Relative Bioavailability of Linaprazan for a New Oral Tablet Formulation of Linaprazan Glurate, and to Assess the Effect of Food on the Pharmacokinetics of Linaprazan
Brief Title: Relative Bioavailability of Linaprazan for the Test Formulation vs. Reference Formulation
Acronym: BA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinclus Pharma Holding AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CX842A2106
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-02

CONDITIONS: Safety; Bioavailability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Reference formulation (Treatment A) (Active Comparator): 100 mg linaprazan glurate reference formulation (4x25 mg oral tablets) in fasting conditions
  Interventions: Drug: Linaprazan glurate
- Test formulation (Treatment B) (Experimental): 100 mg linaprazan glurate test formulation (1x100 mg oral tablet) in fasting conditions
  Interventions: Drug: Linaprazan glurate
- Test Formulation (Treatment C) (Experimental): 100 mg linaprazan glurate test formulation (1x100 mg oral tablet) in fed conditions
  Interventions: Drug: Linaprazan glurate

INTERVENTIONS:
Drug: Linaprazan glurate — 100 mg
  Other Names: formerly X842

SUMMARY:
This is a single-center, open-label, randomized, single dose, 3-way crossover study in healthy volunteers designed to evaluate the relative bioavailability of a new oral tablet formulation of linaprazan glurate in comparison to a previously studied oral tablet formulation under fasting conditions, and to assess the effect of a high fat, high calorie meal on the pharmacokinetics (PK) of linaprazan glurate and the active substance linaprazan after the administration of the new oral tablet formulation.

ELIGIBILITY:
Main Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female aged 18 to 65 years, inclusive.
3. Body mass index ≥18.5 and ≤30.0 kg/m2.
4. Medically healthy, without abnormal clinically significant medical history
5. Female subjects of childbearing potential, as well as their partners and male subjects and their partners, who agree to using methods of contraception
6. Willing and able to consume the high-fat, high calorie breakfast

Exclusion Criteria:

1. Female subjects of childbearing potential unless they agree to use highly effective methods of contraception (failure rate of <1%) from 2 weeks prior to dosing until the end-of-study visit.
2. Male subjects with a partner of childbearing potential, unless they agree to use method of contraception from 2 weeks prior to dosing until the end-of-study visit.History of or current clinically significant disease as defined in the protocol
3. History of or current clinically significant disease as defined in the protocol.
4. History of GERD, significant acid reflux.
5. Subjects who are pregnant, currently breastfeeding, or intend to become pregnant (female subjects) or father a child (male subjects) during the course of the study (i.e., from screening to end of study visit).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS d.o.o., Ljubljana, Ukmarjeva Ulica 6, Slovenia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited form CRS's database of healthy volunteers. All Volunteers were recruited in Slovenia, Ljubljana.
Pre-assignment Details: Approximately 84 healthy volunteers were planned to be screened to achieve 54 randomized subjects. 97 Volunteers were actually screened for eligibility, of those, 67 were Randomized and 49 Analyzed.
Groups:
- Treatment Sequence A B C: Treatments A = 100 mg reference formulation (formulation A) non-fasted B = 100 mg test formulation (formulation B) non-fasted C = 100 mg test formulation (formulation B) fasted
- Treatment Sequence A C B: Treatments A = 100 mg reference formulation (formulation A) non-fasted C = 100 mg test formulation (formulation B) fasted B = 100 mg test formulation (formulation B) non-fasted
- Treatment Sequence B A C: Treatments B = 100 mg test formulation (formulation B) non-fasted A = 100 mg reference formulation (formulation A) non-fasted C = 100 mg test formulation (formulation B) fasted
- Treatment Sequence B C A: Treatments B = 100 mg test formulation (formulation B) non-fasted C = 100 mg test formulation (formulation B) fasted A = 100 mg reference formulation (formulation A) non-fasted
- Treatment Sequence C A B: Treatments
  C = 100 mg test formulation (formulation B) fasted A = 100 mg reference formulation (formulation A) non-fasted B = 100 mg test formulation (formulation B) non-fasted
- Treatment Sequence C B A: Treatment C = 100 mg test formulation (formulation B) fasted B = 100 mg test formulation (formulation B) non-fasted A = 100 mg reference formulation (formulation A) non-fasted
- Exploratory Arm A B C; Exploratory Arm A C B: Subjects underdosed when receiving treatment A, receiving only 1x25 mg LG instead of 4x25. Subjects were excluded from the PK analysis set and their data are instead presented here as exploratory. Treatment sequence as in the title.
Period: Treatment Period 1
Arm/Group | Treatment Sequence A B C | Treatment Sequence A C B | Treatment Sequence B A C | Treatment Sequence B C A | Treatment Sequence C A B | Treatment Sequence C B A | Exploratory Arm A B C | Exploratory Arm A C B
Started (13 subjects were underdosed in treatment period A, receiving 1x25 mg LG instead of 4x25 mg. These 13 subjects completed their remaining treatments but were excluded from the PK analysis set and were therefore given a separate "exploratory arm" when presented here.) | 9 | 9 | 9 | 9 | 9 | 9 | 6 | 7
Completed | 9 | 9 | 7 | 9 | 9 | 8 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 7
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Period: Treatment Period 2
Arm/Group | Treatment Sequence A B C | Treatment Sequence A C B | Treatment Sequence B A C | Treatment Sequence B C A | Treatment Sequence C A B | Treatment Sequence C B A | Exploratory Arm A B C | Exploratory Arm A C B
Started (Treatment period 2 means for example if a subject was randomized to treatment sequence C A B, he/she would receive treatment A in this treatment period.) | 9 | 9 | 7 | 9 | 9 | 8 | 0 | 0
Completed | 7 | 9 | 7 | 9 | 9 | 8 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence A B C | Treatment Sequence A C B | Treatment Sequence B A C | Treatment Sequence B C A | Treatment Sequence C A B | Treatment Sequence C B A | Exploratory Arm A B C | Exploratory Arm A C B
Started (Treatment period 3 means for example if a subject was randomized to treatment sequence C A B, he/she would receive treatment B in this treatment period.) | 7 | 9 | 7 | 9 | 9 | 8 | 0 | 0
Completed | 7 | 9 | 7 | 9 | 9 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 13 subjects were erroneously underdosed with 1x25 mg LG instead of 4x25 mg in the sequence arms starting with treatment A. These 13 subjects were excluded from the analysis set and replaced. Data was collected nevertheless and presented as "exploratory". This is why there is an imbalance between the number in the first two sequence arms.
  In addition, in error, one subject recieved the treatments in reverse order from his/her randomization. E.g. B C A instead of as randomized to A C B.
Groups:
- Treatment Sequence A B C; Treatment A C B; Treatment B A C; Treatment B C A; Treatment C A B; Treatment C B A: Treatments A = 100 mg reference formulation non-fasted B = 100 mg test formualtion non-fasted C = 100 mg test formulation fasted
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A B C | Treatment A C B | Treatment B A C | Treatment B C A | Treatment C A B | Treatment C B A | Total
Number analyzed (Participants) | 15 | 15 | 9 | 10 | 9 | 9 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 9 | 10 | 9 | 9 | 67
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: In error, one subject recieved the treatments in reverse order from what he/she was randomized to. E.g. in the order B C A as opposed to randomized A C B.
  years | 22.2 [19 to 26] | 24.3 [18 to 35] | 26.4 [19 to 45] | 21.5 [18 to 25] | 29.6 [19 to 48] | 22.3 [19 to 26] | 24.1 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 8 | 2 | 6 | 3 | 35
  Male | 8 | 6 | 1 | 8 | 3 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 9 | 10 | 9 | 9 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Slovenia | 15 | 15 | 9 | 10 | 9 | 9 | 67

OUTCOME MEASURES:

1. Primary Outcome: Relative Bioavailability of Linaprazan Comparing Test Formulation vs. Reference Formulation of Linaprazan Glurate. Ratios of AUCinf and AUClast
Description: The Ratio of Area Under the plasma concentration vs. time Curve (AUC) from time 0 to infinity (AUCinf), and from time 0 to last measurement (AUClast) of linaprazan, comparing test formulation vs reference formulation (treatments B vs treatment A) for Relative Bioavailability, i.e. how much linaprazan exposure is increased or decreased with the new formulation.
Time Frame: From pre-dose up to 72 h post dose
Population: PK Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: hours * nmol/Liter
Groups:
- Reference Formulation (Treatment A): 4 x 25 mg linaprazan glurate reference formulation, fasting conditions
- Test Formulation (Treatment B): 100 mg linaprazan glurate test formulation, fasting conditions
  Linaprazan glurate: 100 mg
Arm/Group | Reference Formulation (Treatment A) | Test Formulation (Treatment B)
Number analyzed (Participants) | 51 | 53
hours * nmol/Liter
  AUCinf: number analyzed (Participants) | 40 | 51
  AUCinf | 12341 (1.51) | 25001 (1.32)
  AUClast | 10016.2 (2.78) | 24175.8 (1.34)
Statistical Analysis 1: Comparison: Reference Formulation (Treatment A) vs Test Formulation (Treatment B); The Ratio of geometric mean AUCinf comparing test formulation fasted (treatment B) vs. reference formulation fasted ( treatment A). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other; p < 0.0001, Mixed Models Analysis; Ratio = 1.9954, 95% CI 2-sided [1.8399 to 2.1641] — Treatment B (1x100 mg test formulation) divided by treatment A (4x25 mg reference formulation)
Statistical Analysis 2: Comparison: Reference Formulation (Treatment A) vs Test Formulation (Treatment B); AUClast: Ratio of geometric mean AUClast comparing test formulation fasted (treatment B) vs. reference formulation fasted (treatment A). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other; p < 0.0001, Mixed Models Analysis; Ratio = 2.1250, 95% CI 2-sided [1.9664 to 2.2963] — Treatment B (1x100 mg test formulation) divided by treatment A (4x25 mg reference formulation)

2. Primary Outcome: Relative Bioavailability of Linaprazan Comparing Test Formulation vs. Reference Formulation of Linaprazan Glurate. Ratio of Cmax
Description: The Ratio of Cmax (highest measured concentration) of linaprazan comparing the test formulation vs reference formulation (treatments B vs treatment A) for Relative Bioavailability, i.e. how much linaprazan exposure is increased or decreased with the new formulation.
Time Frame: From pre-dose up to 72 h post dose
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Reference Formulation (Treatment A) | Test Formulation (Treatment B)
Number analyzed (Participants) | 51 | 53
nmol/L | 1430 (1.83) | 3462.2 (1.25)
Statistical Analysis 1: Comparison: Reference Formulation (Treatment A) vs Test Formulation (Treatment B); Ratio of geometric mean Cmax comparing test formulation fasted (treatment B) vs. reference formulation fasted (treatment A). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 2.3167, 95% CI 2-sided [2.0922 to 2.5652] — Treatment B (1x100 mg test formulation) divided by treatment A (4x25 mg reference formulation)

3. Primary Outcome: Relative Bioavailability of Linaprazan Test Formulation in Fed vs. Fasting Conditions, Based on the Means Ratios for AUCinf and AUClast
Description: The Ratio of Area Under the plasma concentration vs. time Curve (AUC) from time 0 to infinity (AUCinf), and from time 0 to last measurement (AUClast) of linaprazan, comparing test formulation vs reference formulation (treatments C vs treatment B) for Relative Bioavailability, i.e. how much linaprazan exposure is increased or decreased in a fed vs fasted state.
Time Frame: From pre-dose up to 72 h post dose
Population: PK Analysis Set.
Measure: Geometric Mean (Standard Deviation); unit: hours * nmol/Liter
Groups:
- Test Formulation (Treatment C): 100 mg linaprazan glurate test formulation, fed conditions
  Linaprazan glurate: 100 mg
Arm/Group | Test Formulation (Treatment B) | Test Formulation (Treatment C)
Number analyzed (Participants) | 53 | 50
hours * nmol/Liter
  AUCinf: number analyzed (Participants) | 53 | 49
  AUCinf | 25001 (1.32) | 19448.9 (1.32)
  AUClast | 24175.8 (1.34) | 19022.8 (1.32)
Statistical Analysis 1: Comparison: Test Formulation (Treatment B) vs Test Formulation (Treatment C); Ratio of geometric mean AUCinf comparing treatment C (fed) versus treatment B (fasted). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 0.7570, 95% CI 2-sided [0.7009 to 0.8177] — Treatment C (1x100 mg test formulation fed) divided by treament B (100 mg test formulation fasted)
Statistical Analysis 2: Comparison: Test Formulation (Treatment B) vs Test Formulation (Treatment C); Ratio of geometric mean AUClast comparing treatment C (fed) versus treatment B (fasted). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 0.7684, 95% CI 2-sided [0.7102 to 0.8313] — Treatment C (1x100 mg test formulation fed) divided by treament B (100 mg test formulation fasted)

4. Primary Outcome: Relative Bioavailability of Linaprazan Test Formulation in Fed vs. Fasting Conditions, Based on the Means Ratios for Cmax
Description: The Ratio of Cmax of linaprazan when comparing test formulation vs reference formulation (treatments C vs treatment B), i.e. how much linaprazan exposure is increased or decreased with the new formulation.
Time Frame: From pre-dose up to 72 h post dose
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Test Formulation (Treatment B) | Test Formulation (Treatment C)
Number analyzed (Participants) | 53 | 50
nmol/L | 3462.2 (1.25) | 1608 (1.29)
Statistical Analysis 1: Comparison: Test Formulation (Treatment B) vs Test Formulation (Treatment C); Ratio of geometric mean Cmax comparing treatment C (fed) versus treatment B (fasted). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 0.2548, 95% CI 2-sided [0.1999 to 0.3247] — Treatment C (1x100 mg test formulation fed) divided by treament B (100 mg test formulation fasted)

5. Secondary Outcome: Relative Bioavailability of Linaprazan Glurate for the Test Formulation vs. Reference Formulation of Linaprazan Glurate, Based on the Means Ratios of PK Parameters.
Description: The Ratio of Area Under the plasma concentration vs. time Curve (AUC) from time 0 to infinity (AUCinf), and from time 0 to last measurement (AUClast) of linaprzan glurate, comparing test formulation vs reference formulation (treatments B vs treatment A) for Relative Bioavailability, i.e. how much linaprazan glurate exposure is increased or decreased with the new formulation.
Time Frame: From pre-dose up to 72 h post dose
Population: PK Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: hours * nmol/Liter
Arm/Group | Reference Formulation (Treatment A) | Test Formulation (Treatment B)
Number analyzed (Participants) | 51 | 53
hours * nmol/Liter
  AUCinf: number analyzed (Participants) | 34 | 41
  AUCinf | 114.2 (1.95) | 320.2 (1.73)
  AUClast | 83.9 (2.49) | 293 (1.84)
Statistical Analysis 1: Comparison: Reference Formulation (Treatment A) vs Test Formulation (Treatment B); Ratio of geometric mean AUCinf comparing test formulation fasted (treatment B) vs. reference formulation fasted ( treatment A). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 3.0245, 95% CI 2-sided [2.5098 to 3.6446] — Treatment B (1x100 mg test formulation) divided by treament A (4x25 mg reference formulation)
Statistical Analysis 2: Comparison: Reference Formulation (Treatment A) vs Test Formulation (Treatment B); Ratio of geometric mean AUClast comparing test formulation fasted (treatment B) vs. reference formulation fasted (treatment A). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 3.5277, 95% CI 2-sided [2.9076 to 4.2799] — Treatment B (1x100 mg test formulation) divided by treament A (4x25 mg reference formulation)

6. Secondary Outcome: Relative Bioavailability of Linaprazan Glurate Comparing Test Formulation vs. Reference Formulation of Linaprazan Glurate. Ratio of Cmax
Description: The Ratio of Cmax (highest measured concentration) of linaprazan glurate comparing the test formulation vs reference formulation (treatments B vs treatment A) for Relative Bioavailability, i.e. how much linaprazan glurate exposure is increased or decreased with the new formulation.
Time Frame: From pre-dose up to 72 h post dose
Population: PK Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Reference Formulation (Treatment A) | Test Formulation (Treatment B)
Number analyzed (Participants) | 51 | 53
nmol/L | 86.8 (2.44) | 214.3 (2.08)
Statistical Analysis 1: Comparison: Reference Formulation (Treatment A) vs Test Formulation (Treatment B); Ratio of geometric mean Cmax comparing test formulation fasted (treatment B) vs. reference formulation fasted ( treatment A). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 3.0245, 95% CI 2-sided [2.5098 to 3.6446] — Treatment B (1x100 mg test formulation) divided by treament A (4x25 mg reference formulation)

7. Secondary Outcome: Relative Bioavailability of Linaprazan Glurate in Fed vs. Fasting Conditions, Based on the Means Ratios for AUCinf, AUClast
Description: The Ratio of Area Under the plasma concentration vs. time Curve (AUC) from time 0 to infinity (AUCinf), and from time 0 to last measurement (AUClast) of linaprazan glurate, comparing test formulation vs reference formulation (treatments C vs treatment B) for Relative Bioavailability, i.e. how much linaprazan glurate exposure is increased or decreased in a fed vs fasted state.
Time Frame: From pre-dose up to 72 h post dose
Population: PK Analysis Set.
Measure: Geometric Mean (Standard Deviation); unit: hours * nmol/Liter
Arm/Group | Test Formulation (Treatment B) | Test Formulation (Treatment C)
Number analyzed (Participants) | 53 | 50
hours * nmol/Liter
  AUCinf: number analyzed (Participants) | 41 | 41
  AUCinf | 320.2 (1.73) | 166.3 (1.52)
  AUClast | 293.0 (1.84) | 144.3 (1.62)
Statistical Analysis 1: Comparison: Test Formulation (Treatment B) vs Test Formulation (Treatment C); [analysis description as in outcome 3, analysis 1]; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 0.4923, 95% CI 2-sided [0.4131 to 0.5867] — Treatment C (1x100 mg test formulation fed) divided by treament B (100 mg test formulation fasted)
Statistical Analysis 2: Comparison: Test Formulation (Treatment B) vs Test Formulation (Treatment C); [analysis description as in outcome 3, analysis 2]; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 0.4923, 95% CI 2-sided [0.4047 to 0.5989] — Treatment C (1x100 mg test formulation fed) divided by treament B (100 mg test formulation fasted)

8. Secondary Outcome: Relative Bioavailability of Linaprazan Glurate in Fed vs. Fasting Conditions, Based on the Means Ratio of Cmax
Description: The Ratio of Cmax of linaprazan glurate when comparing test formulation vs reference formulation (treatments C vs treatment B), i.e. how much linaprazan glurate exposure is increased or decreased with the new formulation.
Time Frame: From pre-dose up to 72 h post dose
Population: PK Analysis Set.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Test Formulation (Treatment B) | Test Formulation (Treatment C)
Number analyzed (Participants) | 53 | 50
nmol/L | 214.3 (2.08) | 55.0 (2.23)
Statistical Analysis 1: Comparison: Test Formulation (Treatment B) vs Test Formulation (Treatment C); Ratio of geometric mean Cmax comparing test formulation fed (treatment C) vs. reference formulation fasted (treatment B). This is a relative comparison, thus there is no unit. The ratio is given under the Estimated value; Test type: Other — Ratio; p < 0.0001, Mixed Models Analysis; Ratio = 0.2522, 95% CI 2-sided [0.1980 to 0.3211] — Treatment C (1x100 mg test formulation fed) divided by treament B (100 mg test formulation fasted)

ADVERSE EVENTS:
Time Frame: Baseline to Visit 5, 1 month
Groups:
- Reference Formulation (Treatment A): 100 mg linaprazan glurate reference formulation (4x25 mg), fasting conditions
  Linaprazan glurate: 100 mg
- Test Formulation (Treatment B): 100 mg linaprazan glurate reference formulation (1x100 mg), fasting conditions
  Linaprazan glurate: 100 mg
- Test Formulation (Treatment C): 100 mg linaprazan glurate test formulation (1x100 mg), fed conditions
  Linaprazan glurate: 100 mg
- Reference: 25 mg linaprazan glurate reference formulation fasting conditions
Arm/Group | Reference Formulation (Treatment A) | Test Formulation (Treatment B) | Test Formulation (Treatment C) | Reference
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/53 | 0/50 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/53 | 0/50 | 0/13
Other Adverse Events (participants affected / at risk) | 17/51 | 12/53 | 14/50 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Formulation (Treatment A) (N=51) | Test Formulation (Treatment B) (N=53) | Test Formulation (Treatment C) (N=50) | Reference (N=13)
Skin Bacterial Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Soft tissue infection with sepsis
OTHER ADVERSE EVENTS (reported when occurring in more than 1.40% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Formulation (Treatment A) (N=51) | Test Formulation (Treatment B) (N=53) | Test Formulation (Treatment C) (N=50) | Reference (N=13)
Tachycardia (Cardiac disorders) | 3 (4) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure diastolic inceased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papula (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vascular disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cardiac disorders (Cardiac disorders) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT05627518/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT05627518/SAP_001.pdf